CLINICAL TRIAL: NCT02868411
Title: Improving the Diagnosis of Traveller's Fevers in Point Of Care (POC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-51; 2012-A01600-43 (Other: ANSM)
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Traveller's Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients admitted for traveller's fever (Experimental)
  Interventions: Other: Rectal Swab

INTERVENTIONS:
Other: Rectal Swab

SUMMARY:
A point-of-care laboratory (POC) was set at North Hospital, Marseille, France for the diagnosis in less than two hours of traveller's fever caused by known pathogens, close to the reception of Emergency service. In this instance 30% of patients have no etiological diagnosis after the POC traveller's fever tests .

The objective of this study is to implement a new diagnosis strategy relying on the hypothesis that a rectal swab would improve the etiological diagnosis of traveller's fever of at least 10%.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted for traveller's fever requiring a microbiological examination with a "Traveller's fever POC kit"
* Patient who freely signed the informed consent form
* Patient affiliated to a social security regime

Exclusion criteria

* Pregnant or breastfeeding women
* Adult patient under guardianship
* Patient deprived with liberty under court order
* Patient refusing or unable to sign the informed consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2013-06-11 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Percentage of patients admitted for traveller's fever with a confirmed etiological diagnosis | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided